# NCT # NCT00318643

# Statistical Analysis Plan

Halozyme Therapeutics, Inc.

Protocol Number: HZ2-05-01

A Phase I-Ha, Multicenter, Open-Label, Multiple Dose, Safety, Tolerability and Pharmacokinetic Study of Recombinant Human Hyaluronidase (Chemophase<sup>TM</sup>) in Combination with Mitomycin in Patients with Non-Muscular-Invasive Bladder Cancer

Sponsor: Halozyme Therapeutics, Inc.

11588 Sorrento Valley Road, Suite 17

San Diego, California 92121

Prepared by:

Synteract, Inc.

5759 Fleet Street, Suite 100

Carlsbad, CA 92008

Version: 4

Date of Creation: September 17, 2006

Last Updated: January 11, 2008

A Phase I-IIa, Multicenter, Open-Label, Multiple Dose, Safety, Tolerability and Pharmacokinetic Study of Recombinant Human Hyaluronidase (Chemophase<sup>TM</sup>) in Combination with Mitomycin in Patients with Non-Muscular-Invasive Bladder Cancer

# **Approval Sheet**

| | Date |
|----------------------------|------|
| alozyme Therapeutics, Inc. | |
| | Date |
| ynteract, Inc. | |

# TABLE OF CONTENTS

| 1. | INTRODUCTION | 4 |
|-----|------------------------------------------------|-----|
| 2. | OBJECTIVES | 4 |
| 3. | STUDY OVERVIEW | 4 |
| 4. | GENERAL ANALYSIS CONSIDERATIONS | 5 |
| 5. | ANALYSIS SETS | |
| 6. | PATIENT DISPOSITION | |
| 7. | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 6 |
| 8. | STUDY DRUG ADMINISTRATION | 6 |
| 9. | PHARMACOKINETIC ANALYSES | 7 |
| 10 | OTHER ANTI CANCER ANALYSES | |
| 11. | SAFETY ANALYSES | 7 |
| | 11.1 Adverse Events | |
| | 11.2 CLINICAL LABORATORY EVALUATION | |
| | 11.3 OTHER SAFETY ANALYSES | 8 |
| | 11.4 CONCOMITANT MEDICATIONS | 9 |
| 12 | LONG-TERM FOLLOW-UP | 9 |
| 13. | SAMPLE SIZE CALCULATION | 9 |
| AP | PENDIX A: LIST OF TABLES, FIGURES AND LISTINGS | 10 |
| AP | PENDIX B: TABLE LAYOUTS | 14 |
| AP | PENDIX C: LISTING LAYOUTS | 56 |
| AP | PENDIX D: INTERNATIONALLY AGREED ORDER FOR SOC | 104 |

3

### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of Halozyme Therapeutics, Inc. Protocol Number HZ2-05-01 [A Phase I-IIa, Open-Label, Multiple Dose, Safety, Tolerability and Pharmacokinetic Study of Recombinant Human Hyaluronidase (Chemophase<sup>TM</sup>) in Combination with Mitomycin in Patients with Non-Muscular-Invasive Bladder Cancer]. The purpose of this plan is to provide specific guidelines from which the analysis will proceed. Any deviations from these guidelines must be substantiated by sound statistical reasoning.

### 2. OBJECTIVES

The primary objectives for this study are the following:

- Determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of escalating doses of Chemophase in combination with mitomycin (Mitomycin, C, MMC) administered as weekly intravesical instillations for five weeks;
- Establish the dose of Chemophase with MMC recommended for future studies.

Secondary objectives for this study include:

- Assess the pharmacokinetics of intravesical administration of MMC alone and in combination with intravesical administration of Chemophase;
- For the patients treated at the MTD, assess the safety and tolerability of intravesical administration of MMC with Chemophase over up to 7 additional maintenance treatments every 3 months following the initial six weekly instillations;
- Observe patients for any preliminary evidence of anti-tumor activity of MMC and Chemophase when combined.

#### 3. STUDY OVERVIEW

This is a Phase I-IIa, open-label, multicenter, dose-escalation, safety, tolerability, and pharmacokinetic study of intravesical treatment with combination of Chemophase and MMC.

Patient may be considered for enrollment in this study if they have initial presentation or recurrence of Stage Ta, T1 or Tis, any grade, bladder cancer after TURBT.

Groups of up to 6 patients will participate in each of the five individual dose cohorts in the dose escalation phase of the study. The amounts of Chemophase to be given for each of the five cohorts are as follows: 20,000 U, 60,000 U, 200,000 U, 400,000 U and 800,000 U. Once the maximum tolerated dose (MTD) has been established, 6 additional

4

evaluable patients will be enrolled at the MTD dose level. This will provide a total of 12 evaluable patients at MTD upon which to confirm safety and tolerability of the MTD regimen. In total, up to 36 evaluable patients will be enrolled. To reach this number, it is anticipated that no more than 44 patients will need to be enrolled.

The MTD will be determined based on number of patients experiencing a dose-limiting toxicity (DLT) at a particular dose level. A patient will be considered to have experienced a DLT if any of the following occur:

- Plasma MMC Concentration >= 100 ng/mL;
- Adverse Event (AE) with a Common Toxicity Criteria (CTC) grade greater than or equal to 3;
- New, treatment-emergent diagnosis of bladder fibrosis.

For further details on MTD determination, refer to the protocol.

Study patients will receive six weekly study treatments followed by post-treatment evaluations, at Weeks 8 and 12. In addition, the twelve patients receiving the MTD will continue to receive combination therapy every 3 months until the end of year 2 or until the time of documented tumor recurrence, whichever occurs first. Long-term follow-up information for those in the MTD cohort will be collected to help make a preliminary assessment of possible anti-tumor activity.

#### 4. GENERAL ANALYSIS CONSIDERATIONS

Statistical analyses will be reported using summary tables, figures, and data listings. No tests for statistical significance will be performed. All analyses and tabulations will be performed using SAS® Version 8.2 on a PC platform. Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentage of patients in corresponding categories. All raw data obtained from the case report forms as well as any derived data will be included in data listings.

#### 5. ANALYSIS SETS

The following patient population sets will be used for analyses:

- The Safety Set will include all patients who received one or more doses of Chemophase. Any patient receiving MMC on study but not receiving Chemophase will be considered for safety, but assessed separately from patients receiving Chemophase for selected analysis;
- The Intent-To-Treat (ITT) Set (for anti-tumor effects) will include all patients receiving one or more doses of Chemophase with MMC. It is recognized that this definition is a modification of the rigid definition of ITT;

5

- The Per-Protocol Set will include all ITT patients who met the following criteria:
  - Satisfied disease-defining Inclusion Criteria #1 and #2;
  - Received at least 4 protocol-specified doses of Chemophase with MMC over an interval not exceeding 8 weeks;
  - o Retained at least 4 intravesical instillations for at least 90 minutes;
  - Were monitored to the time of tumor recurrence, or at least 5 years, whichever occurs first.

Anti-tumor analysis will be performed on the ITT and Per Protocol Sets. In the event all patients in the ITT Set are also in the Per Protocol Set, analysis will only be carried out on the ITT Set.

Baseline and safety analysis will be performed on the Safety Set. Any patient who received MMC on study but not Chemophase will be considered for selected safety assessments; however, those patients will be assessed separately from patients receiving Chemophase.

#### 6. PATIENT DISPOSITION

Patient disposition information will be summarized for all patients. Summaries will include: the number of enrolled patients, the number of patients in each analysis set, the number of patients completing the study without premature withdrawal, and the reasons for not completing the study.

# 7. DEMOGRAPHIC AND BASELINE CHARACTERISTICS

Demographic variables include: age, sex, ethnicity, and race. Other baseline characteristics include: Karnofsky performance status, medical history, urologic history and bladder cancer history. Patient history endpoints to be summarized include the years since initial bladder cancer diagnosis, total number of bladder cancer occurrences, estimated bladder capacity, total number of bladder tumor treatments, total number of bladder cancer surgeries, total number of previous cystoscopies with tumor detected and without tumor detected. When applicable, demographic and baseline characteristics will be summarized.

### 8. STUDY DRUG ADMINISTRATION

For each visit during the study drug administration phase of the study other than Day 1, patients are expected to receive a pre-specified amount of Chemophase, MMC and sterile saline based on the cohort they are assigned to (on Day 1, patients will only receive MMC). Counts and percentages of those patients who receive the pre-specified dose of study drug as well as those who do not will be displayed by cohort and visit. Also summarized will be the instillation dwell time (end time of instillation minus post-instillation void time).

For amount of study drug and sterile saline to be administered for each cohort at each visit, refer to Table 9.3-A of the protocol.

#### 9. PHARMACOKINETIC ANALYSES

The plasma concentrations for MMC and plasma concentrations of rHuPH20 are part of the study design, but will not be summarized in tabular form as part of the analysis plan. Concentrations will be presented in listings.

### 10 OTHER ANTI CANCER ANALYSES

Plasma determinations for rHuPH20 neutralizing antibodies are part of this study design, but will not be summarized in tabular form as part of this analysis plan. Plasma determinations for antibodies will be presented in listings.

All patients completing the study will have a cystoscopy performed at the Week 12 visit. For those patients being treated at MTD, cystoscopies will be performed every three months through the end of Year 2 starting 3 months after the last study drug treatment, which is anticipated to be at Week 6. Endpoints to be collected include the cystoscopy result and the estimated bladder capacity. Summaries of these endpoints will be presented by cohort.

Biomarker tests, consisting of NMP22 BladderChek tests and UroVysion tests, are to be conducted during Week 1 and Week 8 of the study. For those patients treated at MTD, these biomarker tests are also to be performed every 3 months, occurring 6 weeks before each every-three-month clinic visit. Results from these tests will be used to construct a shift table with possible results of positive, negative, no valid result and not done for the BladderChek test and negative, positive, equivocal, other and not done for the Urovysion test.

### 11. SAFETY ANALYSES

All patients who received Chemophase will be included in the safety analyses. Patients who receive MMC, but not Chemophase, will be summarized separately for adverse events. Analysis will consist of point estimates and the 95% confidence interval constructed around the point estimates for the overall incidence of adverse events.

## 11.1 Adverse Events

The adverse events considered are Treatment Emergent Adverse Events (TEAE) defined as those AEs that occurred after initial study drug dosing (first dose of MMC) and those existing AEs that worsened after initial study drug dosing. All listings and tabular summaries of AEs will be restricted to only TEAEs, except for a separate listing showing only those AEs that are pre-treatment-emergent, should any such AEs exist in the

database. Verbatim terms on case report forms will be mapped to preferred terms and system organ classes using the MedDRA dictionary (version 8.0, or a later version at the discretion of Synteract). If a patient has more than one adverse event mapped to the same preferred term, that adverse event will be reported only once in a given summary table using the highest severity and/or closest relationship to study medication. Patient incidence of adverse events will be displayed by system organ class (SOC) and preferred term. Adverse events will also be summarized by severity and relationship to each study drug (Chemophase, MMC) independently. Patient incidence of serious adverse events (including deaths) will also be displayed. Tabular summaries of AEs will list SOCs according to the internationally agreed order, and within each individual SOC the AEs will be listed in order of decreasing incidence. See Appendix D for the internationally agreed order for SOC.

## 11.2 Clinical Laboratory Evaluation

Descriptive statistics of clinical laboratory assessment changes will be presented for baseline and each post baseline time point. In addition, shift tables will be presented to assess abnormal laboratory values over time. In constructing shift tables, baseline results will be compared to the most abnormal post baseline result. Laboratory parameters will be classified as low, normal, high and patient counts of shifts from baseline will be presented. The designation of clinical significance will be displayed.

Listings will be provided for laboratory analyte values. Values outside of the normal range will be flagged as either high or low and the designation of clinical significance will be displayed.

## 11.3 Other Safety Analyses

Complete physical examinations will occur at screening and Week 8. In addition, targeted physical examinations will take place through the study drug administration phase of the study. Shift tables will be created for each body system to show any abnormal result both pre- and post-study drug.

Results for vital signs will be summarized by cohort for each visit. In addition, change from baseline will be presented.

Information for 12-Lead ECG will be collected at screening and Week 8. A shift table of the results for the test will be displayed along with summary statistics of QT, QTc, Heart Rate, P-R Interval and QRS.

The Karnofsky Performance Status will performed on each patient at each visit. Results will be shown by visit and cohort.

#### 11.4 Concomitant Medications

Concomitant medications taken during the time period beginning 28 days prior to initial dosing, on Day 1/Week 1, through the Week 12 assessment (and, for MTD patients continuing on study drug treatment, through the last study drug instillation) will be collected in this study. Concomitant medications will be linked to generic terms and ATC classes using the WHO dictionary, Version 4.3. Concomitant medication use will be presented in listings.

### 12 LONG-TERM FOLLOW-UP

The twelve patients receiving the MTD will continue to receive combination therapy every 3 months until the end of Year 2 or until the time of documented tumor recurrence, whichever occurs first. During this time of extended, long-term, treatment information collected on patients will include vital signs, targeted physical examinations, cystoscopy and urine cytology, urine dipsticks, hematology results, study drug administration, AE collection, concomitant medications and NMP22 BladderChek and UroVysion biomarker tests. Results for endpoints collected will be summarized in similar manner as the regular dosing portion of the study, except results will be presented for only the MTD cohort.

In addition, any patients reported to have tumor recurrences will be recorded. The data will be assessed to make Kaplan Meier estimates of time to tumor recurrence at 6, 12, 18 and 24 months as well as determine median time to tumor recurrence. All other information on tumor recurrences including number of tumors, TNM stage and grading will be shown in listings.

#### 13. SAMPLE SIZE CALCULATION

This is a Phase I-IIa multiple dose study of Chemophase, and is neither designed nor powered for formal statistical comparisons.

# APPENDIX A: LIST OF TABLES, FIGURES AND LISTINGS

# **List of Tables**

| Table | |
|--------|---------------------------------------------------------------------|
| Number | Table Description |
| 1 | Patient Disposition |
| 2 | Demographic Characteristics |
| 3 | Abnormal Medical History at Baseline (Safety) |
| 4 | Urologic History/ Bladder Cancer History |
| 5 | Bladder Treatments/ Surgeries/ Procedures |
| 6 | Study Drug Administration |
| 7 | Cystoscopy at Week 12 |
| 8.1 | NMP22 BladderChek Test |
| 8.2 | UroVysion FISH Biomarker Test |
| 9.1 | Adverse Events by System Organ Class |
| 9.2 | Adverse Events by System Organ Class and Severity |
| 9.3 | Adverse Events by System Organ Class and Relationship to Chemophase |
| 9.4 | Adverse Events by System Organ Class and Relationship to MMC |
| 9.5 | Serious Adverse Events by System Organ Class |
| 10 | Clinical Laboratory Results |
| 11 | Shift Tables of Clinical Laboratory Results |
| 12 | Physical Examination |
| 13 | Vital Signs |
| 14.1 | Shift Table of 12-Lead ECG |
| 14.2 | 12-Lead ECG |
| 15 | Karnofsky Performance Study |
| 16 | Long-Term Follow-Up- Vital Signs |
| 17 | Long-Term Follow-Up- Physical Examination |
| 18 | Long-Term Follow-Up- Cystoscopy |
| 19 | Long-Term Follow-Up- Hematology |
| 20 | Long-Term Follow-Up- Study Drug Administration |
| 21 | Long-Term Follow-Up- NMP22 BladderChek Biomarker Test |
| 22 | Long-Term Follow-Up- UroVysion Biomarker Test |
| 23 | Long-Term Follow-Up- Time to Tumor Recurrence from First Study Drug |
| | Administration (months) |

# **List of Figures**

| Figure<br>Number | Figure Description |
|---|---|
| 1.1 | Time to Tumor Recurrence from First Study Drug (ITT Set) |
| 1.2 | Time to Tumor Recurrence from First Study Drug (Per Protocol Set) (If needed) |

# **List of Data Listings**

| Listing | | <b>CRF Plate</b> |
|---|---|---|
| Number | Listing Description | Number |
| 1 | Patient Disposition | Derived |
| 2 | Inclusion Criteria | 1, 2 |
| 3 | Exclusion Criteria | 3,4 |
| 4 | Criteria Waiver | 5 |
| 5 | Demographics | 6 |
| 6 | Medical History | 7 |
| 7 | Urologic History / Bladder Cancer History | 8 |
| 8 | Previous Bladder Tumor Treatments | 9 |
| 9 | Previous Bladder Surgeries/Cystoscopies with Tumors Detected | 10 |
| 10 | Previous Bladder Cystoscopies without Tumors | 11 |
| 11 | Previous Bladder Fibrosis / Contracture | 12 |
| 12 | Previous Cystometrogram | 12 |
| 13 | Instillation of Chemophase and MMC | 25,26 |
| 14 | Blood Collection and Results for MMC, rHuPH20 and Neutralizing | 27 |
| | Antibodies (NAB) to rHuPH20 | |
| 15 | Urine Cytology | 17 |
| 16 | Cystoscopy | 17 |
| 17 | Urine Dipstick | 23 |
| 18.1 | NMP22 BladderChek Biomarker Test | 24 |
| 18.2 | UroVysion FISH Biomarker Test | 31 |
| 19.1 | Adverse Events (Treatment-Emergent) | 97 |
| 19.2 | Pre-Treatment-Emergent Adverse Events | 97 |
| 20 | Serious Adverse Events | 97 |
| 21 | Reference Range Lab Normals - Hematology | 350 |
| 22 | Reference Range Lab Normals - Chemistry | 351,352 |
| 23 | Reference Range Lab Normals - Urinalysis | 353 |
| 24 | Hematology Results | 19 |
| 25 | Chemistry Results | 20,21 |
| 26 | Urinalysis Results | 22 |
| 27 | Physical Examination | 14,15 |
| 28 | Vital Signs and Karnofsky Performance Status | 13,16 |
| 29 | 12-Lead ECG | 18 |
| 30 | Pregnancy | 18 |
| 31 | Concomitant Medications | 95 |
| 32 | Procedures | 96 |
| 33 | Comments | 98 |
| 34 | Death Report | 101 |
| 35 | Tumor Recurrence | 30 |

| 36 | Long-Term Follow-Up | 28,29 |
|----|------------------------------------------------------------|---------|
| 37 | Utility Database Panel for Dose-Limiting Toxicities (DLTs) | Derived |

**APPENDIX B: TABLE LAYOUTS** 

Table 1
Patient Disposition
All Patients

| | 20,000 U | 60,000 U | 200,000 U | 400,000 U | 800,000 U | Total |
|---|---|---|---|---|---|---|
| Patients Enrolled [1] | n | n | n | n | n | n |
| Received MMC Only | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Safety Set [2] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ITT Set [3] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Per Protocol Set [4] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Completed Study Without Premature Withdrawal | | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Reasons Patient Did Not Complete Study [5] | | | | | | |
| Did not receive all expected instillations of study drug | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Protocol Violation | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Lost to Follow-up | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Non-compliance | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Patient Decision | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Investigator Decision | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Percentage based on number of patients enrolled.

path\t\_program.sas date time

<sup>[1]</sup> Assigned to a treatment cohort.

<sup>[2]</sup> Received at least one dose of Chemophase.

<sup>[3]</sup> Received at least one dose of Chemophase with MMC.

<sup>[4]</sup> Satisfied Inclusion Criteria 1 and 2; received at least 4 doses of Chemophase with MMC over an interval that did not exceed 8 weeks; retained at least 4 intravesical instillations for at least 90 minutes. Note: the criterion "monitored to the time of tumor recurrence, or at least 5 years, whichever occurs first" was not applied for the generation of this table.

<sup>[5]</sup> Patient may have more than one reason for not completing study.

Table 2.1 Demographic Characteristics Safety Set

| | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| A ( ) [1] | . , | | | , | ` , | , , |
| Age (years) [1] | | | | | | |
| n<br>M (GD) | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX |
| Sex | | | | | | |
| Male | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ethnicity | | | | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Race | | | | | | |
| White | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Black, of African Heritage | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| American Indian or Alaska Native | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Multiple Races | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) |
| Combination 1 | m (0/) | n (0/) | m (0/) | ·· (0/) | ·· (0/) | - (0/) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Combination 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

[1] Age is calculated from the date of informed consent. path\t\_program.sas date time

Programmer Note Tables 2.2-2.3 will be for the ITT and Per Protocol Sets (if needed).

Table 3 Abnormal Medical History at Baseline Safety Set

| | 20,000 U | 60,000 U | 200,000 U | 400,000 U | 800,000 U | Total |
|---|---|---|---|---|---|---|
| Body System | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) |
| Respiratory | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cardiovascular | n (%) | 3 2 | n (%) | n (%) | n (%) | |
| Gastrointestinal | | n (%) | | | | n (%) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hepatic | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Endocrine/Metabolic | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Central Nervous System | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hematopoietic/Lymphatic | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dermatological | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Musculoskeletal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Genitourinary/Reproductive | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Psychiatric | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Alcohol/Drug Abuse | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Drug Allergy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Non-Drug Allergy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| HEENT | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Table 4 Urologic History/ Bladder Cancer History Safety Set

| | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Years Since Initial Diagnosis [1] | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Total Number of Bladder Cancer Occurrences | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Most Recent Estimated Bladder Capacity (mL) | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | xx.x |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | XX, XX | xx, xx |

<sup>[1]</sup> Years Since Initial Diagnosis= (Informed Consent Date- Date of Initial Bladder Cancer Diagnosis + 1)/(365.25). path\t\_program.sas date time

Programmer Note: Years Since Initial Diagnosis is calculated as the difference in years between the Date of Initial Bladder Cancer Diagnosis (MHSTDT) and the Date of Informed Consent (IEDT). If only the year of Initial Bladder Cancer Diagnosis is reported then calculate the difference using only the years.

Table 5
Bladder Treatments/ Surgeries/ Procedures
Safety Set

| | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Total Number of Previous Bladder Tumor Treatments [1] | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Total Number of Previous Bladder Surgeries | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Total Number of Previous Cystoscopies With Tumors Detected | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x | xx.x | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Total Number of Previous Cystoscopies Without Tumors Detected | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X | xx.x | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

[1] Each "treatment" may include multiple cycles of the same treatment. path\t\_program.sas date time

Table 6
Study Drug Administration
Safety Set

| Visit | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total (N=) |
|---|---|---|---|---|---|---|
| | (-, / | (2.) | (2.) | (= : ) | (= : ) | (2) |
| Week 1, Day 1 | n | n | n | n | n | n |
| Dose of MMC Instilled | | | | | | |
| 40 mg | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Volume of MMC Instilled | | | | | | |
| 20 mL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dwell Time (min) [1] | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | xx.x | XX.X | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

[1] Dwell Time= (Time of post-instillation voiding- end time of instillation) . path $\t$ \_program.sas date time

Programmer Note Table will repeat for each day study drug is administered.

Table 6 Study Drug Administration Safety Set

| Visit | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Week 2, Day 8 | n | n | n | n | n | n |
| Volume of Chemophase Instilled | | | | | | |
| Expected Volume | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Units of Chemophase Instilled | | | | | | |
| Expected Units | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Volume of Saline Instilled | | | | | | |
| Expected Volume | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dose of MMC Instilled | | | | | | |
| 40 mg | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Volume of MMC Instilled | | | | | | |
| 20 mL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total Volume Instilled | | | | | | |
| 28 mL | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dwell Time (min) [1] | | | | | | |
| N | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

[1] Dwell Time= (Time of post-instillation voiding- end time of instillation) . path \t\_program.sas date time

Programmer Note Table will repeat for each day study drug is administered.

Table 7 Cystoscopy at Week 12 ITT Set

| | 20,000 U | 60,000 U | 200,000 U | 400,000 U | 800,000 U | Total |
|---|---|---|---|---|---|---|
| | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) |
| Result | , | , | | , | , | , |
| | n<br>(0/) | n | n | n | n | n<br>(0/) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Estimated Bladder Capacity Volume | | | | | | |
| n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx xx) | xx.x (xx.xx) | xx x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx x | XX.X | XX.X | xx.x | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Absence of Tumor Recurrence Verified | | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| path\t_program.sas date time | (70) | (/0) | (/0) | (78) | (/%) | -1 (70) |

Programmer Note Table using ITT Set will be renumbered to 7.1 if analysis for Per Protocol Set is needed. Table number for Per Protocol Set will be 7.2.

Table 8.1 NMP22 BladderChek Biomarker Test at Week 8 ITT Set Part 1 of 2

| | | | | | | | | | | Basel | ine [1] | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 20,000 | U (N=) | | | 60,000 | U (N=) | | | 200,000 | ) U (N=) | | | 400,000 | ) U (N=) | | | 800,000 | ) U (N=) | |
| Time Point | Neg | Pos | Inv[2] | ND[3] | Neg | Pos | Inv[2] | ND[3] | Neg | Pos | Inv[2] | ND[3] | Neg | Pos | Inv[2] | ND[3] | Neg | Pos | Inv[2] | ND[3] |
| Week 8 | n | | | | n | | | | n | | | | n | | | | n | | | |
| Negative | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Positive | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No Valid Result (Invalid) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Done | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

If more than one test results is collected, the last repeated test is used.

path\t\_program.sas date time

Programmer Note Table using ITT Set will be renumbered to 8.1.1 if analysis for Per Protocol Set is needed. Table number for Per Protocol Set will be 8.1.2.

<sup>[2]</sup> Inv= No Valid Result (Invalid)

<sup>[3]</sup> ND= Not Done

Table 8.1 NMP22 BladderChek Biomarker Test at Week 8 ITT Set Part 2 of 2

| | | Basel | ine [1] | |
|---------------------------|-------|-------|---------|-------|
| | | Total | (N=) | |
| Time Point | Neg | Pos | Inv[2] | ND[3] |
| Week 8 | n | | | |
| Negative | n (%) | n (%) | n (%) | n (%) |
| Positive | n (%) | n (%) | n (%) | n (%) |
| No Valid Result (Invalid) | n (%) | n (%) | n (%) | n (%) |
| Not Done | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

If more than one test results is collected, the last repeated test is used.

path\t\_program.sas date time

Programmer Note Table using ITT Set will be renumbered to 8.1.1 if analysis for Per Protocol Set is needed. Table number for Per Protocol Set will be 8.1.2.

<sup>[2]</sup> Inv= No Valid Result (Invalid)

<sup>[3]</sup> ND= Not Done

Table 8.2 UroVysion FISH Biomarker Test at Week 8 ITT Set

| | Baseline [1] | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 20 | (1) U 000, | V=) | | | 60 | (1) U 000, | V=) | | | 200 | ),000 U ( | N=) | | | 400 | ,000 U ( | N=) | |
| Time Point | Neg | Pos | Eq[2] | Oth[3] | ND[4] | Neg | Pos | Eq[2] | Oth[3] | ND[4] | Neg | Pos | Eq[2] | Oth[3] | ND[4] | Neg | Pos | Eq[2] | Oth[3] | ND[4] |
| Week 8 | n | | | | | n | | | | | n | | | | | n | | | | |
| Negative | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Positive | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Equivocal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Done | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date

Programmer Note Table using ITT Set will be renumbered to 8.2.1 if analysis for Per Protocol Set is needed. Table number for Per Protocol Set will be 8.2.2.

<sup>[2]</sup> Eq= Equivocal [3] Oth= Other

<sup>[4]</sup> ND= Not Done

Table 8.2 **UroVysion FISH Biomarker Test at Week 8** ITT Set

| | | | | | Baseli | ne [1] | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | 800 | ),000 U ( | N=) | | | - | Γotal (N= | =) | |
| Time Point | Neg | Pos | Eq[2] | Oth[3] | ND[4] | Neg | Pos | Eq[2] | Oth[3] | ND[4] |
| Week 8 | n | | | | | n | | | | |
| Negative | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Positive | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Equivocal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Done | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Programmer Note Table using ITT Set will be renumbered to 8.2.1 if analysis for Per Protocol Set is needed. Table number for Per Protocol Set will be 8.2.2.

<sup>[2]</sup> Eq= Equivocal [3] Oth= Other

<sup>[4]</sup> ND= Not Done

Table 9.1 Treatment Emergent Adverse Events by System Organ Class [1] Safety Set

| System Organ Class / Preferred Term | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total [2]<br>(N=) | Received Only MMC (N=) |
|---|---|---|---|---|---|---|---|
| Patients Experiencing at Least One Adverse<br>Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 95% CI [3] | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | $(xx \ x, xx \ x)$ | (xx.x, xx.x) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once.

path\t\_program.sas date time

<sup>[2]</sup> Total column does not consider patients that received only MMC.
[3] 95% Confidence Interval based on a binomial distribution.

Table 9.2

Treatment Emergent Adverse Events by System Organ Class and Severity [1]

Safety Set
Part 1 of 2

| | 2 | 0,000 U (N= | =) | 6 | 0,000 U (N | =) | 20 | 00,000 U (N | I=) | 40 | 00,000 U (N | (=) | 80 | 00,000 U (N | (=) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Mild | Mod | Sev | Mild | Mod | Sev | Mild | Mod | Sev | Mild | Mod | Sev | Mild | Mod | Sev |
| Patients Experiencing at Least One Adverse<br>Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

[1] At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once using the highest severity. path\t\_program.sas date time

Table 9.2 Treatment Emergent Adverse Events by System Organ Class and Severity [1]
Safety Set
Part 2 of 2

| | | Total (N=) | 1 |
|---|---|---|---|
| System Organ Class / Preferred Term | Mild | Mod | Sev |
| Patients Experiencing at Least One Adverse<br>Event | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once using the highest severity. path\t\_program.sas date

Table 9.3 Treatment Emergent Adverse Events by System Organ Class and Relationship to Chemophase [1] Safety Set

| | 20,000 | U (N=) | 60,000 | U (N=) | 200,000 | U (N=) | 400,000 | U (N=) | 800,000 | ) U (N=) | Total | (N=) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] |
| Patients Experiencing at Least One Adverse<br>Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once using the closest relationship to Chemophase.
[2] Includes all events reported as "Possibly", "Probably", or "Related" relationship to Chemophase.

path\t\_program.sas date time

<sup>[3]</sup> Includes all events reported as "Unlikely", or "Not Related" relationship to Chemophase.

Table 9.4 Treatment Emergent Adverse Events by System Organ Class and Relationship to MMC [1] Safety Set

| | 20,000 | U (N=) | 60,000 | U (N=) | 200,000 | ) U (N=) | 400,000 | U (N=) | 800,000 | ) U (N=) | Total | (N=) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] | Related [2] | Not Rel [3] |
| Patients Experiencing at Least One Adverse<br>Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 . | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once using the closest relationship to MMC. [2] Includes all events reported as "Possibly", "Probably", or "Related" relationship to MMC.

<sup>[3]</sup> Includes all events reported as "Unlikely", or "Not Related" relationship to MMC.

path\t\_program.sas date time

Table 9.5 Treatment Emergent Serious Adverse Events by System Organ Class [1] Safety Set

| System Organ Class / Preferred Term | 20,000 U<br>(N=) | 60,000 U<br>(N=) | 200,000 U<br>(N=) | 400,000 U<br>(N=) | 800,000 U<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Patients Experiencing at Least One Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

.

path\t\_program.sas date time

<sup>[1]</sup> At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once.

**Table 10.1 Clinical Laboratory Results: Hematology** Safety Set WBC (unit)

| | 20,000 U (N=) | | 60,000 U (N=) | | 200,000 U (N=) | | 400,000 | ) U (N=) | 800,000 | ) U (N=) | Total (N=) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | | | | | |
| n | n | | n | | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | xx, xx | | XX, XX | | XX, XX | | XX, XX | | xx, xx | | XX, XX | |
| Above Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Below Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Week 2, Day 8 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Above Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Below Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration. [2] Change= Change from Baseline

path\t\_program.sas date

Table will repeat for each analyte for each time point.

Programmer note In most cases, baseline will be Week 1, Day 1.

**Table 10.2** Clinical Laboratory Results : Chemistry Safety Set Sodium (unit)

| | 20,000 | U (N=) | 60,000 U (N=) | | 200,000 U (N=) | | 400,000 | ) U (N=) | 800,000 | U (N=) | Total (N=) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | | | | | |
| n | n | | n | | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | XX.X | | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | | xx, xx | | xx, xx | | xx, xx | |
| Above Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Below Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Week 2, Day 8 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Above Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Below Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration. [2] Change= Change from Baseline

path\t\_program.sas date

Table will repeat for each analyte for each time point.

Programmer note In most cases, baseline will be Week 1, Day 1.

**Table 10.3** Clinical Laboratory Results : Urinalysis Safety Set Specific Gravity

| | 20,000 U (N=) | | 60,000 U (N=) | | 200,000 U (N=) | | 400,000 | ) U (N=) | 800,000 | U (N=) | Total (N=) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | | | | | |
| n | n | | n | | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | XX.X | | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | | xx, xx | | xx, xx | | xx, xx | |
| Above Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Below Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Week 2, Day 8 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Above Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Below Normal | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration. [2] Change= Change from Baseline

path\t\_program.sas date

Table will repeat for each analyte for each time point.

Programmer note In most cases, baseline will be Week 1, Day 1.

**Table 11.1** Shift Tables of Clinical Laboratory Results : Hematology Safety Set Part 1 of 2

| | Baseline [1] | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 20,000 U (N=) | | | 60,000 U (N=) | | | 200,000 U (N=) | | | 400,000 U (N=) | | | 800,000 U (N=) | | |
| Most Abnormal Post Baseline Result [2] | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| WBC (unit) | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ANC (unit) | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| RBC (unit) | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Table will repeat for each analyte.

Programmer note In most cases, baseline will be Week 1, Day 1.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] A patient will be assigned a "High" score for post baseline result if a patient has both a high and low post baseline result.
**Table 11.1** Shift Tables of Clinical Laboratory Results : Hematology Safety Set Part 2 of 2

| | | Baseline [1 | 1 |
|----------------------------------------|-------|-------------|-------|
| | | Total (N=) | |
| Most Abnormal Post Baseline Result [2] | High | Normal | Low |
| WBC (unit) | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |
| ANC (unit) | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |
| RBC (unit) | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |
| ••• | | | |
| ••• | | | |

path\t\_program.sas date time

Table will repeat for each analyte.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] A patient will be assigned a "High" score for post baseline result if a patient has both a high and low post baseline result.

Table 11.2 Shift Tables of Clinical Laboratory Results : Chemistry Safety Set Part 1 of 2

| | | | | | | | | Baseline [1 | ] | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 2 | 0,000 U (N: | =) | 6 | 0,000 U (N | =) | 20 | 00,000 U (N | (=) | 40 | 00,000 U (N | I=) | 80 | 00,000 U (N | (=) |
| Most Abnormal Post Baseline Result [2] | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| Sodium (unit) | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Potassium (unit) | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Chloride (unit) | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

• • •

path\t\_program.sas date time

Table will repeat for each analyte.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

<sup>[2]</sup> A patient will be assigned a "High" score for post baseline result if a patient has both a high and low post baseline result.

Table 11.2 Shift Tables of Clinical Laboratory Results : Chemistry Safety Set Part 2 of 2

| | | Baseline [1] | |
|----------------------------------------|-------|--------------|-------|
| | | Total (N=) | |
| Most Abnormal Post Baseline Result [2] | High | Normal | Low |
| Sodium (unit) | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |
| Potassium (unit) | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |
| Chloride (unit) | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| | ` / | ` / | ` / |
| Low | n (%) | n (%) | n (%) |

...

path\t\_program.sas date time

Table will repeat for each analyte.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

<sup>[2]</sup> A patient will be assigned a "High" score for post baseline result if a patient has both a high and low post baseline result.

**Table 11.3** Shift Tables of Clinical Laboratory Results: Urinalysis Safety Set Part 1 of 2

| | | | | | | | | Baseline [1] | ] | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 2 | 0,000 U (N= | =) | 6 | 0,000 U (N= | =) | 20 | 00,000 U (N | [=) | 40 | 00,000 U (N | =) | 80 | 00,000 U (N | =) |
| Most Abnormal Post Baseline Result [2] | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low | High | Normal | Low |
| Specific Gravity | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| рН | n | | | n | | | n | | | n | | | n | | |
| High | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

 $path \\ t\_program.sas \quad date$ time

Programmer note In most cases, baseline will be Week 1, Day 1. Also, only those analytes with numeric results will be considered.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] A patient will be assigned a "High" score for post baseline result if a patient has both a high and low post baseline result.

**Table 11.3** Shift Tables of Clinical Laboratory Results: Urinalysis Safety Set Part 2 of 2

| | | Baseline [1] | |
|----------------------------------------|-------|--------------|-------|
| | | Total (N=) | |
| Most Abnormal Post Baseline Result [2] | High | Normal | Low |
| S : C C : | | | |
| Specific Gravity | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |
| рН | n | | |
| High | n (%) | n (%) | n (%) |
| Normal | n (%) | n (%) | n (%) |
| Low | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Programmer note In most cases, baseline will be Week 1, Day 1. Also, only those analytes with numeric results will be considered.

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] A patient will be assigned a "High" score for post baseline result if a patient has both a high and low post baseline result.

Table 12 Physical Examination [1] Safety Set

| | | | | | | Pr | e-Study Drug | 5 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 20,000 | ) U (N=) | 60,00 | 0 U (N=) | 200,000 | ) U (N=) | 400,000 | 0 U (N=) | 800,00 | 0 U (N=) | Tota | 1 (N=) |
| Post-Study Drug | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal | Normal | Abnormal |
| Respiratory | n | | n | | n | | n | | n | | n | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cardiovascular | n | | n | | n | | n | | n | | n | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Gastrointestinal | n | | n | | n | | n | | n | | n | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> For both pre- and post baseline results, a patient is considered normal for body system unless a result of abnormal is reported for specified body system and time interval.

Table 13 Vital Signs Safety Set Heart Rate (unit)

| | 20,000 | U (N=) | 60,000 | U (N=) | 200,000 | U (N=) | 400,000 | ) U (N=) | 800,000 | ) U (N=) | Total | l (N=) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | | | | | |
| n | n | | n | | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | xx, xx | | XX, XX | | XX, XX | | xx, xx | | xx, xx | | xx, xx | |
| Week 2, Day 8 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| Week 3, Day 15 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx |
| | ••• | | | | | ••• | | | | | ••• | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Table will repeat for each vital sign at each time point.

<sup>[2]</sup> Change= Change from Baseline

**Table 14.1** Shift Table of 12-Lead ECG Safety Set Part 1 of 2

| | | | | | | | | Screening | 5 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 20 | 0,000 U (N | I=) | 60 | 0,000 U (N | [=) | 20 | 0,000 U (N | V=) | 40 | 0,000 U (N | V=) | 80 | 0,000 U (N | <b>1</b> =) |
| Week 8, Day 50 | Nor[1] | Abn[2] | ACS[3] | Nor[1] | Abn[2] | ACS[3] | Nor[1] | Abn[2] | ACS[3] | Nor[1] | Abn[2] | ACS[3] | Nor[1] | Abn[2] | ACS[3] |
| | | | | | | | | | | | | | | | · |
| | n | | | n | | | n | | | n | | | n | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

[1] Nor= Normal

[2] Abn= Abnormal, not Clinically Significant [3] ACS= Abnormal, Clinically Significant

**Table 14.1** Shift Table of 12-Lead ECG Safety Set Part 2 of 2

| | | Screening Total (N=) | |
|---|---|---|---|
| Week 8, Day 50 | Nor[1] | Abn[2] | ACS[3] |
| | n | (0/) | (0/) |
| Normal | n (%)<br>n (%) | n (%)<br>n (%) | n (%)<br>n (%) |
| Abnormal, not Clinically Significant<br>Abnormal, Clinically Significant | n (%) | n (%) | n (%) |

- [1] Nor= Normal
- [2] Abn= Abnormal, not Clinically Significant [3] ACS= Abnormal, Clinically Significant

Table 14.2 12-Lead ECG Safety Set

| | 20,000 | U (N=) | 60,000 | U (N=) | 200,000 | U (N=) | 400,000 | ) U (N=) | 800,000 | U (N=) | Total | l (N=) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Result | Change [1] | Result | Change [1] | Result | Change [1] | Result | Change [1] | Result | Change [1] | Result | Change [1] |
| QT (unit) | | | | | | | | | | | | |
| Screening | | | | | | | | | | | | |
| n | n | | n | | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | | xx, xx | | xx, xx | | xx, xx | |
| Week 8, Day 50 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| QTc (unit)<br>Screening | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

[1] Change= Change from Baseline

path\t\_program.sas date time

Table will repeat for each ECG parameter.

Table 15 **Karnofsky Performance Status** Safety Set

| | 20,000 | U (N=) | 60,000 | U (N=) | 200,000 | U (N=) | 400,000 | ) U (N=) | 800,000 | ) U (N=) | Total | l (N=) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] | Result | Change [2] |
| Baseline [1] | | | | | | | | | | | | |
| n | n | | n | | n | | n | | n | | n | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | XX, XX | | xx, xx | | xx, xx | | XX, XX | |
| 100% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 90% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 80% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 70% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 60% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 50% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 40% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 30% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 20% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 10% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| 0% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |
| Week 2, Day 8 | | | | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| 100% | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | | n (%) | |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.
[2] Change= Change from Baseline

path\t\_program.sas date time

Table will repeat for each available time point.

Programmer note In most cases, baseline will be Week 1, Day 1. Categories may collapsed as requested by client.

Table 16 Long-Term Follow-Up- Vital Signs Safety Set Heart Rate (unit)

| | MTD Cohort (N=) | |
|--------------|-----------------|--------------|
| | Result | Change [2] |
| Baseline [1] | | |
| n | n | |
| Mean (SD) | xx.x (xx.xx) | |
| Median | XX.X | |
| Min, Max | XX, XX | |
| Month 4 ½ | | |
| n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX |
| Month 7 ½ | | |
| n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x |
| Min, Max | XX, XX | xx, xx |
| | | ••• |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Table will repeat for each vital sign parameter for each long-term follow-up time point.

Programmer note In most cases, baseline will be Week 1, Day 1 and should exactly match baseline expressed in table 13 (Vital Signs).

<sup>[2]</sup> Change= Change from Baseline

Table 17 Long-Term Follow-Up- Targeted Physical Examination Safety Set

| | MTD Cohort |
|---|---|
| Reported at least one instance of abnormality [1]: | (N=) |
| Pre-Study Drug | |
| | (0/) |
| Respiratory | n (%) |
| Cardiovascular | n (%) |
| Gastrointestinal | n (%) |
| Hepatic | n (%) |
| Post-Study Drug up to and including Week 12 Visit | |
| Respiratory | n (%) |
| Cardiovascular | n (%) |
| Gastrointestinal | n (%) |
| Hepatic | n (%) |
| Post-Study Drug during Long-Term Follow-Up Starting with Month 6 until Study Discontinuation | |
| Respiratory | n (%) |
| Cardiovascular | n (%) |
| Gastrointestinal | n (%) |
| Hepatic | n (%) |
| | ( / • / ) |

Patients reporting more than one abnormality for the same system will be only counted once per time period (pre-study drug/ post-study drug).

path\t\_program.sas date time

Programmer note The first two endpoints should match up exactly with first two endpoints on table 12 (Physical Examination)

#### Table 18 Long-Term Follow-Up- Cystoscopy ITT Set Month 4 ½

| | MTD Cohort<br>(N=) |
|----------------------------------------|--------------------|
| Cystoscopy | |
| Result | |
| Normal | n (%) |
| Abnormal, Not Clinically Significant | n (%) |
| Abnormal, Clinically Significant | n (%) |
| Estimated Bladder Capacity Volume (mL) | |
| n | n |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| Min, Max | XX, XX |
| ••• | |

path\t\_program.sas date time

Repeat table for each time point.

Table 19 Long-Term Follow-Up- Hematology Safety Set WBC (unit)

| | MTD Cohort (N=) | |
|--------------|-----------------|--------------|
| | Result | Change [2] |
| Baseline [1] | | |
| n | n | |
| Mean (SD) | xx.x (xx.xx) | |
| Median | xx.x | |
| Min, Max | XX, XX | |
| Month 4 ½ | | |
| n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx |
| Month 7 ½ | | |
| n | n | n |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx |

<sup>[1]</sup> Baseline defined as measurement taken most closely prior to first study drug administration.

path\t\_program.sas date time

Table will repeat for each analyte for each long-term follow-up time point.

Programmer note In most cases, baseline will be Week 1, Day 1 and should exactly match baseline expressed in table 10.1 (Hematology Results).

<sup>[2]</sup> Change= Change from Baseline

Table 20 Long-Term Follow-Up- Study Drug Administration Safety Set

| /isit | MTD Cohort<br>(N=) |
|---------------------------------------------------------|--------------------|
| Month 4 ½ | |
| Chemophase | |
| Units Instilled- Mean (SD) | xx.x (xx.xx) |
| Volume Instilled- Mean (SD) | xx.x (xx.xx) |
| Sterile Saline | |
| Volume Instilled- Mean (SD) | xx.x (xx.xx) |
| MMC | |
| Dose Instilled- Mean (SD) | xx.x (xx.xx) |
| Volume Instilled- Mean (SD) | xx.x (xx.xx) |
| Total Volume Instilled- Mean (SD) | xx.x (xx.xx) |
| Any Interruptions or Adjustments Due to DLTs? | |
| Yes | n (%) |
| No | n (%) |
| Length of Time Patient Retain Solution in their Bladder | |
| 2 Hours | n (%) |
| >= 90 Minutes, < 2 Hours | n (%) |
| < 90 Minutes | n (%) |
| 5 mL Urine Sample Collected and Frozen? | |
| Yes | n (%) |
| No | n (%) |

path\t\_program.sas date time

Table will repeat for each analyte for each long-term follow-up time point.

Table 21 Long-Term Follow-Up- NMP22 BladderChek Biomarker Test Safety Set

| | MTD Cohort<br>(N=xx) |
|-----------------|----------------------|
| Manuals 2 | |
| Month 3 | |
| Negative | n (%) |
| Positive | n (%) |
| No Valid Result | n (%) |
| Not Done | n (%) |
| Month 6 | |
| Negative | n (%) |
| Positive | n (%) |
| No Valid Result | n (%) |
| Not Done | n (%) |

...

path\t\_program.sas date time

Table will repeat for each analyte for each long-term follow-up time point.

Table 22 Long-Term Follow-Up- UroVysion FISH Biomarker Test Safety Set

| | MTD Cohort<br>(N=xx) |
|-----------|----------------------|
| 4.42 | |
| Month 3 | |
| Negative | n (%) |
| Positive | n (%) |
| Equivocal | n (%) |
| Other | n (%) |
| Not Done | n (%) |
| Month 6 | |
| Negative | n (%) |
| Positive | n (%) |
| Equivocal | n (%) |
| Other | n (%) |
| Not Done | n (%) |

path\t\_program.sas date time

Table will repeat for each analyte for each long-term follow-up time point.

Table 23
Long-Term Follow-Up- Time to Tumor Recurrence from First Study Drug Administration (Months)
Safety Set

| | MTD Cohort |
|----------------------------------------|---------------|
| Category, n (%) | (N=xx) |
| Number Patients with Tumor Recurrence | n |
| Number Patients Censored | n |
| Quartiles (95% CI): | |
| 25 <sup>th</sup> Percentile | x.x(x.x, x.x) |
| 50 <sup>th</sup> Percentile (median) | x.x(x.x, x,x) |
| 75 <sup>th</sup> Percentile | x.x(x.x, x.x) |
| Kaplan Meier Estimate (# at Risk) | |
| 6 Months | x.x (n) |
| 12 Months | x.x (n) |
| 18 Months | x.x (n) |
| 24 Months | x.x (n) |
| Range (Patients with Tumor Recurrence) | xx, xx |
| Range (All Patients) | XX, XX |

#### **APPENDIX C: LISTING LAYOUTS**

### Listing 1 Patient Disposition (N=)

| Cohort X/ | | | Safety | | Per Protocol | Date of Study Discontinuation/ | Completed | Reason for | Date of Investigator's | Name of |
|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units P | Patient ID Re | ceived MMC Only? | Set [1] | ITT Set [2] | Set [3] | Study Termination | Study? | Discontinuation [4] | Signature | Investigator |

[1] Received at least one dose of Chemophase.

<sup>[2]</sup> Received at least one dose of Chemophase with MMC.

<sup>[3]</sup> Satisfied Inclusion Criteria 1 and 2; received at least 4 doses of Chemophase with MMC over an interval that did not exceed 8 weeks; retained at least 4 intravesical instillations for at least 90 minutes. Note: the criterion "monitored to the time of tumor recurrence, or at least 5 years, whichever occurs first" was not applied for the generation of this table.

<sup>[4]</sup> Reasons for discontinuation include: Did not receive all expected instillations of study drug. Protocol Violation, Lost to Follow-up, Adverse Event, Non-compliance, Patient Decision, Investigator Decision, Other.

#### Listing 2 Inclusion Criteria (N=)

| Cohort X/ | Patient | Date Informed | | Inclusion Criteria | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Consent Signed | 1a | 1b | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |

path\t\_program.sas date time

Programmer Note Inclusion criteria to be shown on separate page.

## Listing 3 Exclusion Criteria (N=)

| Cohort X/ | | Date Informed | | Exclusion Criteria | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | Patient ID | Consent Signed | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |

path\t\_program.sas date time

Programmer Note Exclusion criteria to be shown on separate page.

#### Listing 4 Criteria Waiver (N=)

| Cohort X/ | Patient | Patient Comply with All | | | If No, Criteria Not Met | | |
|---|---|---|---|---|---|---|---|
| Chem Units | ID | Entry Criteria? | Criteria Not Met | Criteria Number | Exemption Explanation | Exemption Granted By | Date of Exemption |
| | | | Inclusion/Exclusion | | | | |

## Listing 5 Demographics (N=)

| Cohort X/ | Patient | | | | | | |
|---|---|---|---|---|---|---|---|
| Chem Units | ID | Date of Birth | Day 1 Dose | Age on Day 1 | Sex | Ethnicity | Race |

#### Listing 6 Medical History (N=)

| Cohort X/ | Patient | Mark if No Medical | | | | |
|---|---|---|---|---|---|---|
| Chem Units | ID | History | Site / System | Description | Year of Diagnosis / Onset | Ongoing |

# Listing 7 Urologic History / Bladder Cancer History Part 1 of 3 (Cancer Recurrences) (N=)

| Cohort X/ Patient | Bladder C | Cancer |
|-------------------|---------------------------|---------------------|
| Chem Units ID | Date of Initial Diagnosis | Date of Recurrences |

#### Listing 7 Urologic History / Bladder Cancer History Part 2 of 3 (Estimation of Bladder Capacity) (N=)

| Cohort X/ | Patient | Bladder Capacity | | |
|---|---|---|---|---|
| Chem Units | ID | Date of Estimation | Method of Estimation | Volume (mL) |

#### Listing 7 Urologic History / Bladder Cancer History Part 3 of 3 (Bladder Symptoms) (N=)

| | _ | Frequent Urination? | | Nighttime Urinations? | | Urinary Urgency? | | Urinary Incontinence? | | Use Pads? | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | | Average | | Average | | Average | | Average | | Average |
| Chem Units | ID | Yes/No | Urinations/Day | Yes/No | Urinations/Night | Yes/No | Urinations/Week | Yes/No | Urinations/Week | Yes/No | Pads/Day |

### Listing 8 Previous Bladder Tumor Treatments (N=)

| Cohort X/ Patient | | Start Date / | | | |
|---|---|---|---|---|---|
| Chem Units ID | Medication / Treatment | Stop Date | Dose / Units | Route | Toxicities |

# Listing 9 Previous Bladder Surgeries / Cystoscopies with Tumors Detected Part 1 of 2 (N=)

| | | | | | Procedure | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | | Tumor # from | | | Tumor Size | Histological | | |
| Chem Units | ID | Mark if None | CRF | Date | Type | (mm) | Grading | Location | TNM Staging |
| | | | | | Surgery | | | | |
| | | | | | Cystoscopy | | | | |

# Listing 9 Previous Bladder Surgeries / Cystoscopies with Tumors Detected Part 2 of 2 (N=)

| Cohort X/ | Patient | | Tumor # from | | If Yes, | | |
|---|---|---|---|---|---|---|---|
| Chem Units | ID | Mark if None | CRF | Biopsy Performed? | Biopsy Findings | Gross Appearance of Tumor | Mucosa or Not Applicable |

### Listing 10 Previous Bladder Cystoscopies without Tumors (N=)

| Cohort X/ | Patient | Mark if | | | |
|---|---|---|---|---|---|
| Chem Units | ID | None | Cystoscopy # from CRF | Date of Procedure | Abnormal Findings |

## Listing 11 Previous Bladder Fibrosis / Contracture (N=)

| Cohort X/ | Patient | Mark if | | | |
|------------|---------|---------|------|-----------|----------|
| Chem Units | ID | None | Date | Diagnosis | Etiology |

## Listing 12 Previous Cystometrogram (N=)

| Cohort X/ | Patient | Mark if | | | | If Abnormal, |
|---|---|---|---|---|---|---|
| Chem Units | ID | None | Test Date | Result | Test(s) Used | Specify Abnormality |

# Listing 13 Instillation of Chemophase and MMC Page 1 of 2 (N=)

| | | Refrain From Drinking Fluids? | | Pre-Instillation | | Instillation | | | Post-Instillation | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | For $\geq = 8$ Hours | During | Fully | Volume Obtained by | | Start | End | Elapsed Time | Time of | Dwell Time | Voided |
| Chem Units | ID | Before Instillation | Instillation | Voided Before? | Catheter (mL) | Date | Time | Time | (min) [1] | Voiding | (min) [2] | Volume (mL) |

[1] Elapsed Time= End Time of Instillation – Start Time of Instillation [2] Dwell Time= Time of Voiding – End Time of Instillation
# Listing 13 Instillation of Chemophase and MMC Page 2 of 2 (N=)

| | | | | Saline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Chemophas | e Instilled | Instilled | MMC Ir | stilled | | | | | |
| Cohort X/ | Patient | Volume | Units | Volume | Volume | Dose | Total Volume | Interrupt/ Adjust | | Time Solution | Post Drug Instillation |
| Chem Units | ID | (mL) | (U) | (mL) | (mL) | (mg) | Instilled (mL) | due to DLTs? | If Yes, Specify | Retained [1] | Urine Sample Collected? |

[1] Possible responses for Time Solution Retained include: 2 Hours, 90 Minutes to <2 Hours, <90 Minutes path\t\_program.sas date time

# Listing 14 Blood Collection and Results for MMC, rHuPH20 and Neutralizing Antibodies (NAB) to rHuPH20 (N=)

| | | | _ | | Collection | | | esults | Neutralizing |
|---|---|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | | Mark if | | | | MMC (ng/mL) | | Antibodies (NAB) to |
| Chem Units | ID | Visit # | Not Done | Date Drawn | Scheduled Time | Actual Time | or Not Done | rHuPH20 (U/mL) | rHuPH20 |

### Listing 15 Urine Cytology (N=)

| | Cohort X/<br>Chem Units | Patient<br>ID | Visit # | Mark if Not<br>Done | Collection Date | Diagnosis | Microscopic Description |
|---|---|---|---|---|---|---|---|
| _ | | | | | | | |

> Listing 16 Cystoscopy (N=)

| Cohort X/ | Patient | | Mark if | Cystoscopy | | If Abnormal, Specify | | Absence of Bladder Cancer |
|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Visit# | Not Done | Date | Result | Abnormality: | Estimated Bladder Capacity (mL) | Verified? |

### Listing 17 Urine Dipstick (N=)

| | _ | Cohort X/<br>Chem Units | Patient<br>ID | Visit<br># | Mark if Not<br>Done | Collection Date | Collection Time | Do Results Indicate Possible UTI? |
|---|---|---|---|---|---|---|---|---|
| | _ | | | | | | | |
| path\t_program.sas | date | time | | | | | | |

### Listing 18.1 NMP22 BladderChek Biomarker Test (N=)

| Cohort X/ | Patient | | Mark if | | | | | |
|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Visit # | Not Done | Test | Collection Date | Collection Time | Result | If Invalid, Was Test Repeated? |
| • | | | | | | | | |

path\t\_program.sas date time

Programmer Note Test column will indicate whether test conducted is an initial test or a retest.

### Listing 18.2 UroVysion FISH Biomarker Test (N=)

| Cohort X/ | Patient | | Mark if Not | | | | |
|---|---|---|---|---|---|---|---|
| Chem Units | ID | Visit # | Done | Test | Collection Date | Collection Time | Result |

path\t\_program.sas date time

Programmer Note Test column will indicate whether test conducted is an initial test or a retest.

#### Listing 19.1 Adverse Events (Treatment-Emergent) (N=)

| | | | | | | | | | Action | Taken with: | Relati | onship to: | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Mark | | | | | | - | | | | | | |
| Cohort X/ | Patient | if | | Preferred Term/ | Start | Stop | Serious | Severity | | | | | | |
| Chem Units | ID | None | AE# | Verbatim Term | Date | Date | ? | (CTC) | MMC | Chemophase | MMC | Chemophase | Other Action | Outcome |

path\t\_program.sas date time

Programmer Note Abbreviations may be needed for some of the columns. If so, add a footnote to define the abbreviations.

<sup>\*</sup> Treatment-Emergent Adverse Events are defined as those adverse events that occurred after initial study drug dosing and those existing AE's that worsened after initial study drug dosing. Adverse Events that occurred after the first dose of MMC but prior to first dose of Chemophase will be indicated with a "\*".

# Listing 19.2 Pre-Treatment-Emergent Adverse Events (N=)

| | | | | | | | | _ | Action | Taken with: | Relati | onship to: | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | Mark<br>if | | Preferred Term/ | Start | Ston | Serious | Severity | | | | | | |
| Chem Units | ID | None | AE# | Verbatim Term | Date | Stop<br>Date | ? | (CTC) | MMC | Chemophase | MMC | Chemophase | Other Action | Outcome |

<sup>\*</sup> Only Adverse Events that occurred between the time the patient signed the informed consent and prior to the first dose of MMC and Chemophase are included.

path\t\_program.sas date time

Programmer Note Abbreviations may be needed for some of the columns. If so, add a footnote to define the abbreviations.

#### Listing 20 Serious Adverse Events (Treatment-Emergent) (N=)

| | | | | | | | | _ | Action | Taken with: | Relati | onship to: | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Mark | | | | | | - | | | | | | |
| Cohort X/ | Patient | if | | Preferred Term/ | Start | Stop | Serious | Severity | | | | | | |
| Chem Units | ID | None | AE# | Verbatim Term | Date | Date | ? | (CTC) | MMC | Chemophase | MMC | Chemophase | Other Action | Outcor |

path\t\_program.sas date time

Programmer Note Abbreviations may be needed for some of the columns. If so, add a footnote to define the abbreviations.

<sup>\*</sup> Treatment-Emergent Adverse Events are defined as those adverse events that occurred after initial study drug dosing and those existing AE's that worsened after initial study drug dosing. Adverse Events that occurred prior to first dose of MMC but prior to first dose of Chemophase will be indicated with a "\*".

### Listing 21 Reference Range Lab Normals – Hematology

| | | | <u>-</u> | Age | | Lab (Both or Male) | | Lab (Female) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site ID | Lab ID | Date<br>Effective | Lab Test | Low | High | Low | High | Low | High | Units |

 $path \\ t\_program.sas \quad date \qquad time$ 

Programmer Note Order the lab tests in the same order as on the CRF.

### Listing 22 Reference Range Lab Normals – Chemistry

| | | <u>-</u> | Age | | Lab (Both or Male) | | Lab (Female) | | |
|---|---|---|---|---|---|---|---|---|---|
| Site ID | Date<br>Effective | Lab Test | Low | High | Low | High | Low | High | Units |
| COVANCE | | | | - | | - | | | |

path\t\_program.sas date time

Programmer Note Order the lab tests in the same order as on the CRF.

### Listing 23 Reference Range Lab Normals – Urinalysis

| | | | | | A | .ge | Lab (Bot | th or Male) | Lab (I | Female) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Site ID | Test<br>Code | Lab<br>Test | Occu<br>Seq | Date Effective | Low | High | Low | High | Low | High | Units |
| COVANCE | | | | | | | | | | | _ |

path\t\_program.sas date time

Programmer Note Order the lab tests in the same order as on the CRF.

### Listing 24 Hematology Results (N=)

| Cohort X/ | Patient | | | | Mark if Not | Collection | Collection | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Lab Test | Visit # | Lab ID | Done | Date | Time | Result [1] | Unit | Abnormal, not CS | Abnormal and CS |

CS = Clinically Significant.

[1] H indicates a value above the normal range. L indicates a value below the normal range.

path\t\_program.sas date time

Programmer Note Put an "H" next to results that are above the normal range. Put an "L" next to results that are below the normal range. Sort the lab tests in the same order as on the CRF.

### Listing 25 Chemistry Results (N=)

| Cohort X/ | Patient | | | | Mark if Not | Collection | Collection | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Lab Test | Visit# | Lab ID | Done | Date | Time | Result [1] | Unit | Abnormal, not CS | Abnormal and CS |
| | | | | COVANCE | | | | | | | _ |

CS = Clinically Significant.

[1] H indicates a value above the normal range. L indicates a value below the normal range.

path\t\_program.sas date time

Programmer Note Put an "H" next to results that are above the normal range. Put an "L" next to results that are below the normal range. Sort the lab tests in the same order as on the CRF.

### Listing 26 Urinalysis Results (N=)

| Cohort X/ | Patient | | | Visit | | Mark if | Collection | Collection | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Lab ID | Lab Test | # | Lab ID | Not Done | Date | Time | Result [1] | Unit | Abnormal, not CS | Abnormal and CS |
| | | | | | COVANCE | | | | | | | |

CS = Clinically Significant.

[1] H indicates a value above the normal range. L indicates a value below the normal range.

path\t\_program.sas date time

Programmer Note Put an "H" next to results that are above the normal range. Put an "L" next to results that are below the normal range. Sort the lab tests in the same order as on the CRF.

## Listing 27 Physical Examination (N=)

| Cohort X/ | Patient | | Mark if | Exam | New, Changed or | PE | | | |
|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Visit # | Not Done | Date | Resolved Abnormality? | # | System | Description of Abnormality | Clinically Significant? |

path\t\_program.sas date time

Programmer Note For System', add footnotes to explain abbreviations as needed.

If Physical Exam was not done, put "Not Done" for Exam Date'.

Sort System by System code #.

# Listing 28 Vital Signs and Karnofsky Performance Status (N=)

| | | | | | | | Blood | Pressure | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | (mı | mHg) | To | emperatu | re | Wei | ght | Hei | ght | |
| | | | Mark if | Date of | | | | | | | | | | | | |
| Cohort X/ | Patient | Visit | Not | Vital | Heart Rate | Respiration | | | | | Coll. | | | | | Karnofsky |
| Chem Units | i ID | # | Done | Collected | (bpm) | (breaths/min) | Systolic | Diastolic | Result | Unit | Type | Result | Units | Result | Units | Score |
| | | | | | | | | | | | Oral | | | | | |
| | | | | | | | | | | | Aural | | | | | |

path\t\_program.sas date time

Programmer Note If vitals were not done put "Not Done" for Date.

> Listing 29 12-Lead ECG (N=)

| Cohort X/ | Patient | | Mark if | ECG | | If Abnormal, CS, | QT | QTc | HR | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Visit # | Not Done | Date | Result | Specify: | (msec) | (msec) | (bpm) | P-R Interval (msec) | QRS (msec) |

> Listing 30 Pregnancy (N=)

| Cohort X/ | Patient | | Mark if | | | |
|---|---|---|---|---|---|---|
| Chem Units | ID | Visit # | Not Done | Date | Reason, If Not Done | Result |

### Listing 31 Concomitant Medications (N=)

| Cohort X/ | Patient | Mark if | Con | | | | | | Date of | | | | Given for | If Yes, AE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | None | Med# | Medication | Dose | Unit | Route | Regimen | Day 1 | Start Date | Stop Date | Indication | AE? | #s |

path\t\_program.sas date time

Programmer Note If there are no concomitant medications put "NONE" for Medication'.

Add footnotes to explain abbreviations as needed.

### Listing 32 Procedures (N=)

| Cohort X/ | Patient | Mark if | Procedure | | | | Related to | If Yes, |
|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | None | # | Procedure | Date | Findings / Results | AE? | AE #s |

path\t\_program.sas date time

Programmer Note If there are no procedures put "NONE" for Procedure'.

### Listing 33 Comments (N=)

| Cohort X/ | Patient | Mark if | | Pertains to Visi | t | |
|---|---|---|---|---|---|---|
| Chem Units | ID | None | Comment # | Date | CRF Page | Comment |

path\t\_program.sas date time

Programmer Note If there are no comments put "NONE" for Comment #'.

# Listing 34 Death Report (N=)

| Cohort X/ | Patient | Date of | Date Death | | Autopsy | | Investigator | |
|---|---|---|---|---|---|---|---|---|
| Chem Units | ID | Death | Reported to Site | Primary Cause | Performed? | Comments | Signed? | Date of Signature |

### Listing 35 Tumor Recurrence (N=)

| | | | | | | | | | | If Yes, | Gross | Involvement of |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | Mark if | Procedure | Procedure | Tumor Size | Histopathological | Tumor | TNM | Biopsy | Biopsy | Appearance | Bladder |
| Chem Units | ID | None | Date | Type | (mm) | Grading | Location | Staging | Performed? | Findings | of Tumor | Mucosa, or NA |

### Listing 36 Long-Term Follow-Up Part 1 of 5 (N=)

| | | | | | | | Bladd | er Cancer T | reatments | |
|---|---|---|---|---|---|---|---|---|---|---|
| Cohort X/<br>Chem Units | Patient<br>ID | Contact/<br>Visit Date | Method of<br>Contact | Patient<br>Status at<br>Contact | Source of Information | Treatment | Mark if<br>None | Start<br>Date | Stop<br>Date | Ongoing? |

### Listing 36 Long-Term Follow-Up Part 2 of 5 (N=)

| | | | | NMP22 BladderChek Test | |
|---|---|---|---|---|---|
| Cohort X/ | Patient | Contact/ Visit | Mark if | Collection | |
| Chem Units | ID | Date | None | Date/Time | Result |

### Listing 36 Long-Term Follow-Up Part 3 of 5 (N=)

| | | | Ţ | UroVysion FISH Biomarker Test | |
|---|---|---|---|---|---|
| Cohort X/ | Patient | Contact/ Visit | Mark if | Collection | |
| Chem Units | ID | Date | None | Date/Time | Result |

### Listing 36 Long-Term Follow-Up Part 4 of 5 (N=)

| | | | | C | ystoscopy | | | Ur | ine Cytologies | S | | Bladder Bio | ppsies |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | If Abnormal, | | | | | | | |
| Cohort X/ | | Contact/ | Mark if | | | Specify | Mark if | | | Microscopic | Mark if | | |
| Chem Units | Patient ID | Visit Date | None | Date | Result | Abnormality | None | Date | Diagnosis | Description | None | Date | Findings |

### Listing 36 Long-Term Follow-Up Part 5 of 5 (N=)

| | | | Tumor Recurrence | | |
|---|---|---|---|---|---|
| Cohort X/<br>Chem Units | Patient ID | Contact/<br>Visit Date | Mark if None | Date Confirmed | Investigator Signed? |

## Listing 37 Utility Database Panel for Dose-Limiting Toxicities (DLTs) (N=)

| | | | | Adverse Event Considered | PK Lab Assessment of | Treatment | |
|---|---|---|---|---|---|---|---|
| Cohort X/ | Patient | Mark if | Date | to be DLT? If so, Name | MMC Level Considered | Emergent Bladder | Reason Given for Discontinuation on |
| Chem Units | ID | No DLT | Reported | Adverse Event | to be DLT? | Fibrosis? | Termination Page |

Protocol defined DLTs are AEs with a CTC grade greater than or equal to 3, Plasma MMC Concentration >=100 ug/mL and Diagnosis of treatment-emergent bladder fibrosis.

### APPENDIX D: INTERNATIONALLY AGREED ORDER FOR SOC

Infections and infestations

Neoplasms benign and malignant (including cysts and polyps)

Blood and the lymphatic system disorders

Immune system disorders

Endocrine disorders

Metabolism and nutrition disorders

Psychiatric disorders

Nervous system disorders

Eye disorders

Ear and labyrinth disorders

Cardiac disorders

Vascular disorders

Respiratory, thoracic and mediastinal disorders

Gastrointestinal disorders

Hepato-biliary disorders

Skin and subcutaneous tissue disorders

Musculoskeletal, connective tissue and bone disorders

Renal and urinary disorders

Pregnancy, puerperium and perinatal conditions

Reproductive system and breast disorders

Congenital and familial/genetic disorders

General disorders and administration site conditions

Investigations

Injury and poisoning

Surgical and medical procedures

Social circumstances

This list is from an EMEA Guideline, 'A Guideline on Summary of Product Characteristics', October 2005.

A Phase I-IIa, Multicenter, Open-Label, Multiple Dose, Safety, Tolerability and Pharmacokinetic Study of Recombinant Human Hyaluronidase (Chemophase<sup>TM</sup>) in Combination with Mitomycin in Patients with Non-Muscular-Invasive Bladder Cancer

### Approval Sheet

| 1/31/08 | Halozyme Therapeutics, Inc. | | 1 (7 )08 |
|-----------------|-----------------------------|-----|-----------------|
| Synteract, Inc. | | · · | 1/31/08<br>Date |